CLINICAL TRIAL: NCT04332250
Title: Influence Of Incomplete Revascularization on Long-Term Outcomes After Primary Percutaneous Coronary Intervention (PPCI). A Single Center Real-Life Retrospective Analysis
Brief Title: Influence Of Incomplete Revascularization on Long-Term Outcomes After Primary Percutaneous Coronary Intervention (PPCI)
Status: Completed | Type: Observational
Sponsor: Amany Edward Ramzy (Other)
Responsible Party: Sponsor-Investigator, Amany Edward Ramzy, Principle investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Amany Edward Ramzy
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Primary Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
evaluate the influence of incomplete revascularization during the index hospitalization on in-hospital and long-term outcomes in STEMI patients undergoing PPCI in Assiut University heart hospital.

DETAILED DESCRIPTION:
* Study groups: Patients will be divided into 2 groups

  1. Group I: Complete revascularization was achieved by PPCI.
  2. Group II: Complete revascularization was not achieved by PPCI.
* In hospital outcomes: All the patients will be reviewed for during hospital admission to record major acute cardiac events (MACE). Only the most serious event of major adverse cardiac events will be used to calculate the cumulative major adverse cardiac events per patient according to the following sequence: (death > heart failure > recurrent non-fatal MI > serious secondary arrhythmia necessitating DC shock> recurrent or refractory angina. MACE will be reported according to the standard definitions.(Tsai IT, et al.,2017)
* Long-term follow-up: The patients will be followed by telephone interviews for all-cause mortality, re-hospitalization by ACS, re-hospitalization by heart failure, planned and unplanned PCI or CABG. Long-term MACE will include: all-cause mortality, re-hospitalization by ACS, re-hospitalization by heart failure, unplanned revascularization. Patients who undergo planned revascularization later on after discharge will be followed till the date of revascularization for actual events and will be censored in Kaplan Meier Survival analysis. These patients will be included in a third group of staged late complete revascularization to be followed for the long-term MACE events starting from the planned revascularization procedure.

ELIGIBILITY:
Inclusion Criteria:

All Patients aged >18 years with STEMI admitted to Assiut University Heart hospital and underwent successful PPCI between January 2016 to December 2019 were recruited. Selection of patients for primary PCI was as per guideline recommendations.

-

Exclusion Criteria:

* Patients with incomplete data.
* Patients with previous coronary artery bypass grafting (CABG).
* Patients presenting with cardiogenic shock, cardiac arrest or pulmonary edema.
* Mechanical complications of MI; namely VSD, wall rupture, mitral regurgitation secondary to papillary muscle or chordal rupture.
* Patients with unsuccessful PPCI with a final TIMI flow ≤ I in infarct related artery.
* Patients with a significant co-morbidity reducing life expectancy to <1 year as patients with advanced liver diseases, cerebrovascular diseases, malignancy and chronic lung diseases that could affect patient prognosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All Patients aged >18 years with STEMI admitted to Assiut University Heart hospital and underwent successful PPCI between January 2016 to December 2019 were recruited. Selection of patients for primary PCI was as per guideline recommendations
Sampling Method: Probability Sample
Enrollment: 3200 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Mace | between January 2016 to December 2019 were recruited
  All the patients will be reviewed for during hospital admission to record major acute cardiac events (MACE). Only the most serious event of major adverse cardiac events will be used to calculate the cumulative major adverse cardiac events per patient according to the following sequence: (death > heart failure > recurrent non-fatal MI > serious secondary arrhythmia necessitating DC shock> recurrent or refractory angina. MACE will be reported according to the standard definitions